CLINICAL TRIAL: NCT03456492
Title: Hyponatremia in Elderly Patients With Fractures Around the Hip; Role of Glutamate (CSF Glutamate Study)
Brief Title: Hyponatremia in Elderly Patients With Fractures Around the Hip.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshymaa Hassan Mohammed, Doctor, Assiut University
Other Study IDs: Hyponatremia in elderly
Record Dates: First submitted 2018-02-13; First posted 2018-03-07 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Hyponatremia in Elderly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- case: Hyponatremic elderly patients (>70 years) with hip fractures
  Interventions: Diagnostic Test: serum sodium
- control: Normonatremic elderly patients(>70 years) undergoing joint replacement
  Interventions: Diagnostic Test: serum sodium

INTERVENTIONS:
Diagnostic Test: serum sodium — Serum sodium will be measured on admission, assesment of mental status by Modified Mini-Mental score and measurement of glutamate in CSF sample taken while dripling during spinal anathesia for surgical intervention.
  Other Names: 3M score; CSF glutamate

SUMMARY:
Hyponatremia was defined as a serum sodium concentration <135 mmol/L that occurred at least once during a patient's hospital stay from admission to discharge. Elderly patients with fragility fractures are particularly susceptible to hyponatremia because of their impaired physiology, multiple comorbidities (such as hypocortisolism, hypothyroidism, hepatic cirrhosis, renal disease, and congestive heart failure), polypharmacy (e.g., antihypertensives, antidepressants, and antiepileptics), hospitalization, perioperative fluid restrictions, and homeostatic stress from the fracture itself and the subsequent surgery.

The study has 2 parts:

Part 1: aims to to find incidence of hyponatremia in sample of 70 elderly patients with fractures around the hip, effect of hyponatremia on mental state of the patients by using Modified Mini-Mental state (3MS) examination and to find mortality rate for 6 months post admission.

Part 2: aims to compare sample of 18 elderly hyponatremic patients with fractures around the hip (case group) with sample of 10 elderly normonatremic patients with osteoartharitis of knee or hip who admitted for elective joint replacement (control group) as regards; serum sodium, 3M score, and CSF glutamate to find correlation between the cognitive status assessed by 3M score and CSF glutamate as a biomarker for hyponatremia.

DETAILED DESCRIPTION:
These patients are also at a higher risk of the complications of hyponatremia such as brain injury, the main result of acute symptomatic hyponatremia and associated with significant morbidity and mortality. Severe hyponatremia (i.e., a serum sodium concentration <125 mmol/L) ), if unrecognized in its first stages and left untreated, has a high rate of mortality; for this reason, an accurate clinical assessment must be made, focusing on fluid status, examining the potential etiology, and conducting the appropriate investigations. In approximately 50% of patients, chronic hyponatremia results from inappropriate antidiuretic hormone secretion. Chronic mild hyponatremia is usually asymptomatic and is traditionally regarded as benign. However, it is associated with a lower bone mineral content and density in nearly all regions of the hip, with more pronounced losses in the trochanteric and femoral neck regions. It can also lead to osteoporosis, abnormal gait patterns, cognitive impairment, bone demineralization, respiratory failure, noncardiogenic pulmonary edema, falls, and fractures. Compared to normonatremic individuals, hyponatremic individuals are known to have a longer time from admission to surgery.

Glutamate which is the main excitatory neurotransmitter in our body may play role in implication of hyponatremia on the brain. Cerebrospinal fluid (CSF) sample can be taken while dripling during spinal anathesia for surgical intervention for determination of glutamate

ELIGIBILITY:
Inclusion Criteria:

* Hyponatremic elderly patients > 70 years with hip fractures (case group) and surgical intervention will be done by spinal anesthesia so; a sample of CSF can be taken.
* Normonatremic elderly patients > 70 years undergoing undergoing joint replacement (control group) and surgical intervention will be done by spinal anesthesia so; a sample of CSF can be taken.

Exclusion Criteria:

* Age < 70 years
* Patients receive general anesthesia.

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly patients > 70 years
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
To find correlation between the cognitive status assessed by 3M score and CSF glutamate as a biomarker for hyponatremia. | baseline

SECONDARY OUTCOMES:
Early diagnosis and treatment of hyponatremia to avoid fractures | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emad Zarief Kamel, MD, Study Chair — Associate professor of anesthesiology and ICU; Mohammed Ismail Sedek, MD, Study Chair — Associate professor of clinical pathology
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Management of hyponatraemia in older people: old threats and new opportunities — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4110800/
- See also: what causes hyponatremia in elderly patients? — http://www.medscape.com/viewarticle/714108
- See also: Prevalence of Hyponatremia in Elderly Patients with Hip Fractures: A Two-Year Study — http://www.ncbi.nlm.nih.gov/pubmed/28810258